CLINICAL TRIAL: NCT06247566
Title: CXCR4-targeted 68Ga-Pentixafor PET/CT for Guiding Surgical Treatment of Primary Aldosteronism With Bilateral Adrenal Lesions: Preliminary Results From a Single-center Retrospective Study
Brief Title: 68Ga-Pentixafor PET/CT for Guiding Surgical Treatment of Primary Aldosteronism With Bilateral Adrenal Lesions
Status: Completed | Type: Observational
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, zhiwei shu, Principal Investigator, Central South University
Other Study IDs: zshu
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Primary Aldosteronism With Bilateral Adrenal Lesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 68Ga-Pentixafor PET/CT: Patients with Primary Aldosteronism (PA) accompanied by bilateral adrenal lesions undergoing 68Ga-Pentixafor PET/CT to discriminate PA forms with unilateral from bilateral excess aldosterone production, so as to determine whether to choose surgical treatment.

SUMMARY:
Screening potential candidates who may benefit from surgery remains challenging for patients diagnosed with primary aldosteronism (PA) accompanied by bilateral adrenal lesions. Although adrenal venous sampling is currently the gold standard, it is a technically cumbersome, challenging, and difficult-to-interpret invasive procedure that requires a cutting-edge facility and radiologists with a high level of expertise, which restricts its widespread use. The present study aimed to assess the comprehensive effect of 68Ga-pentixafor positron emission tomography/computer tomography (PET/CT) on guiding surgical treatments for PA patients with bilateral adrenal lesions.

DETAILED DESCRIPTION:
Primary aldosteronism (PA) is characterized by the overproduction of renin-independent aldosterone, which results in increased blood volume, potassium excretion, and sodium storage in the body, as well as the inhibition of renin-angiotensin system activity. Clinically, the condition frequently presents as hypertension and hypokalemia. Patients with PA are at a much higher risk of experiencing cardiovascular and cerebrovascular complications than those with primary hypertension matched by blood pressure. PA is classified into two subtypes: unilateral aldosterone hypersecretion (most often aldosterone-producing adenoma (APA)) and contralateral aldosterone non-secretion or bilateral aldosterone hypersecretion (most often idiopathic hyperaldosteronism (IHA)). Differentiating PA subtypes is crucial, as patients with unilateral adrenal hypersecretion of aldosterone may be cured by the surgical removal of the adrenal lesion. Moreover, mineralocorticoid-receptor antagonists (MRAs) are the choice therapy for patients with bilateral hypersecretion.

Computed tomography (CT) is a useful tool for identifying and analyzing abnormalities in the adrenal gland and is one of the main methods used to distinguish between unilateral and bilateral adrenal lesions. CT images with abnormalities on only one side of the adrenal gland in young PA patients (aged <35 years) suggest that abnormal hypersecretion of aldosterone is caused by the unilateral adrenal lesion. However, PA patients with bilateral adrenal lesions on CT do not necessarily exhibit excessive aldosterone secretion. Aldosterone hypersecretion may occur in only one side of the gland. However, because CT does not provide enough information about the secretory activity of a detected nodule, it is difficult to distinguish the side of the adrenal lesion that secretes excessive aldosterone. In recent years, adrenal vein sampling (AVS) - which determines lesions with functional aldosterone secretion - has been considered the gold standard for identifying PA subtypes with bilateral adrenal lesions. However, the feasibility of AVS remains controversial because of its substantial cost, invasiveness with potential risks, and complicated technique with a relatively high rate of failure. Therefore, in regions where AVS is infeasible, experienced physicians may recommend MRAs treatment directly, or the suspected aldosterone-producing lesions may be removed based on the severity of the disease and adrenal CT features. In the latter setting, larger lesions or the side of lesions with radiological features of classic cortical adenoma are often removed, but these lesions may be non-functional. Therefore, this empirical method has a high risk of failure in disease control. Hence, considerable efforts have been made to identify a cost-effective, convenient, and non-invasive substitution for AVS. The utilization of functional imaging techniques is promising for detecting aldosterone-secreting adrenal lesions. For instance, the performance of 11C-metomidate positron emission tomography/computer tomography (PET/CT) is comparable to that of AVS. However, the short half-life of 11C-metomidate and higher requirements for equipment limits its widespread application in clinical practice.

The C-X-C chemokine receptor 4 (CXCR4) - a G protein-coupled transmembrane receptor - is highly expressed in aldosterone-producing tissue16. Its expression is strongly correlated with the expression of aldosterone synthase CYP11B2 (cytochrome P450, family, subfamily b, polypeptide 2). The utilization of 68Ga-pentixafor, a radiolabeled CXCR4 ligand, enables the visualization of tissues exhibiting elevated CXCR4 expression on PET/CT by specifically binding to CXCR4 receptors on the cell membrane 18. Evidence has shown that the utilization of 68Ga-pentixafor PET/CT in patients with adrenal lesions reveals a notable disparity in the uptake value of the tracer between the adrenal lesion side generating excessive aldosterone and non-functional adrenal adenomas (NFA). Previous study also showed that 68Ga-pentixafor PET/CT has diagnostic significance in PA subtypes. We found that the maximum standardized uptake value (SUVmax) of IHA lesions and NFA was significantly lower than that of APA. However, studies on the value of PET/CT in patients with PA coupled with bilateral adrenal lesions are scanty. Herein, we employed 68Ga-pentixafor PET/CT imaging to evaluate PA patients with bilateral adrenal lesions who may receive surgical benefits and tracked their prognosis to examine the significance of 68Ga-pentixafor PET/CT in guiding the treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

patients with bilateral adrenal lesions who were diagnosed as PA

Exclusion Criteria:

1. patients diagnosed with other types of secondary hypertension
2. patients had comorbidities
3. Patients with incomplete follow-up data
4. Patients who successfully underwent AVS

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with bilateral adrenal lesions who were diagnosed as PA from January 1, 2020, to July 1, 2023
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
the the maximum standardized uptake value of adrenal lesions | January 1st 2021 - July 1st 2023

SECONDARY OUTCOMES:
number of patients with lateralization indicated by PET/ CT | January 1st 2021 - July 1st 2023
number of the patients undergoing adrenalectomy | January 1st 2021 - July 1st 2023

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Xiangya Hospital, Central South University, Changsha, Hu'nan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shu Z, He Y, Long T, Guo M, Xia Z, Fu X, Li B, Zhang B, Yang Y, Chen J, Jiang T, Chen X, Cheng K, Liu L, Gan Y. Is CXCR4-targeted 68Ga-pentixafor PET/CT a reliable AVS-free modality for surgical decision-making and prognostic prediction in primary aldosteronism with bilateral adrenal lesions? EJNMMI Res. 2025 Aug 28;15(1):111. doi: 10.1186/s13550-025-01309-4. PMID 40875090